CLINICAL TRIAL: NCT05804825
Title: Message Testing Protocol for Misinformation Concerns
Brief Title: Testing the Persuasiveness of Pro-inoculation Arguments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: dfjgehea
Record Dates: First submitted 2022-10-20; First posted 2023-04-07 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Vaccination Hesitancy; Human Papillomavirus Vaccination; Vaccine Refusal
Keywords: misinformation; HPV vaccine; vaccine hesitancy
MeSH Terms: conditions — Vaccination Hesitancy; Vaccination Refusal; Communication

STUDY DESIGN:
Intervention Model Description: randomized discrete choice modeling experiment design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simple forewarning message (Active Comparator): Participants will receive a simple short forewarning message to read and rate.
  Interventions: Behavioral: Simple forewarning message
- Argument inoculation messages (Experimental): Participants will view a random sample of 3 text-only short messages (from a corpus of 100 arguments) to read and rate.
  Interventions: Behavioral: Argument inoculation messages

INTERVENTIONS:
Behavioral: Argument inoculation messages — Participants will then be presented with arguments randomly selected by the Qualtrics software algorithm from the full set of messages.
  Arms: Argument inoculation messages
Behavioral: Simple forewarning message — Participants will be presented with a simple forewarning message.
  Arms: Simple forewarning message

SUMMARY:
The investigators will recruit a national sample of parents of 7-10-year-olds to complete an argument strength ranking for either a simple forwarding message or between 3 and 6 randomly selected arguments from an overall set of 50 to 100 messages identified from various online sources. Parents will rate each message they see on measures of perceived argument strength/PME. Parents will also answer sociodemographic questions and then rank the believability of a set of anti-vaccine messages identified in a different study. Study findings will contribute valuable information to understanding the effectiveness of different inoculation messages.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female parent or legal guardian of an adolescent ages 7-10
2. Age eligible child has not yet received any doses of the HPV vaccine
3. Resides in the United States
4. English speaking
5. Completed informed consent

Exclusion Criteria:

1. Unable to read English at a 6th grade literacy level
2. Age < 18
3. Does not have a child within the age range of 7-10
4. Age-eligible child has received 1 or more doses of the HPV vaccine
5. Does not have a social media account on one or more of the following platforms OR does not read online news stories: Twitter, Instagram, YouTube, Facebook (feasibility testing only - survey participation will not have this exclusion criteria)
6. Unwilling or unable to provide informed consent to study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 523 (Actual)
Dates: Start 2023-05-04 (Actual); Primary Completion 2023-05-24 (Actual); Study Completion 2023-05-24 (Actual)

PRIMARY OUTCOMES:
Argument strength/PME | The outcome measure will be assessed immediately after the participant has viewed each pro-HPV vaccine message if they are in the multiple message condition, or the simple message if they are in the simple message condition stimuli during the survey.
  Arguments will be rated for their argument strength/message effectiveness
Misinformation believability | The outcome measure will be assessed immediately after the participant has viewed each misinformation message during the survey.
  A rating of the believability/ credibility of vaccine misinformation

CONTACTS AND LOCATIONS:
Locations (1):
- UPenn, Philadelphia, Pennsylvania, United States